CLINICAL TRIAL: NCT03156387
Title: Patient Perceptions and Clinical Efficacy of Frenectomies Using Diode Laser Versus Conventional Techniques
Brief Title: Clinical Efficacy of Frenectomies Using Diode Laser Versus Conventional Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: T.C. Dumlupınar Üniversitesi (Other)
Responsible Party: Principal Investigator, Berceste Guler, Clinical Investigator, T.C. Dumlupınar Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-KAEK-86/05
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: High Frenum Attachment
Keywords: diode laser; scalpel surgery; frenectomy; postoperative complications
MeSH Terms: conditions — Postoperative Complications | interventions — Lasers, Semiconductor; Laser Therapy

STUDY DESIGN:
Intervention Model Description: This study, designed as a randomized prospective controlled clinical trial, was conducted to compare the clinical outcomes of frenectomies performed using conventional surgery or a diode laser.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diode laser (Experimental): A 2.8 W, 980 nm diode laser(Sirona Advanced) in continuous wave mode with an air cooling handpiece was used in the alternative frenectomy technique. The frenulum was held with a hemostat, and a repeated continuous wave mode was applied for the excision. It was also used to remove the periosteal adhesion. The remnants of the ablated tissue were removed with saline, and no sutures were placed after the diode laser treatment.
  Interventions: Procedure: Diode laser
- Scalpel (Active Comparator): (1) topical anesthesia (20% benzocaine), (2) local anesthesia using the bilateral vestibular infiltration technique, with 0.6 ml (1/3 of the carpule contents) of 4% articaine and 1:200,000 epinephrine, (3) hemostatic clamping of the frenulum, (4) excision of the whole band of tissue, together with its alveolar attachment, with a 15C scalpel blade, (5) relaxation and unbending of any fibrous adhesions to the underlying periosteum, and (6) simple suturing with 5-0 silk thread
  Interventions: Procedure: Scalpel

INTERVENTIONS:
Procedure: Diode laser — 2.8 W diode laser surgery were applied on high frenulum attachment and follow-up VAS scores were evaluated
  Other Names: Sirona Advanced
  Arms: Diode laser
Procedure: Scalpel — Scalpel surgery were performed after local anesthetic administration and VAS scores were recorded.
  Arms: Scalpel

SUMMARY:
The aim of present study was to compare the keratinized gingival tissue measurements, degree of subjective complaints, and functional complications of using an 980 nm diode laser versus a scalpel for frenectomies. Thirty-six patients requiring frenectomies, between 18 and 51 years old, were randomly assigned to either scalpel or diode laser treatments. The soft tissue measurements, including the keratinized gingiva width (KGW), attached gingiva width(AGW), and attached gingiva thickness (AGT), were recorded before surgery, immediately after, one week later, and one, three, and six months after surgery. In addition, the functional complications and the morbidity (level of pain, swelling, and redness) were evaluated during the first postoperative week using a visual analog scale (VAS). The VAS scores indicated that the patients treated with a diode laser had less discomfort and functional complications compare with scalpel surgery.

DETAILED DESCRIPTION:
The whole mouth records of each participant served as a basis for the clinical periodontal diagnoses. Prior to the frenectomy, the same investigator recorded the following parameters: plaque index (PLI), gingival index (GI), pocket probing depth (PD), clinical attachment level (CAL), and bleeding on probing (BOP). All of the clinical parameters were measured at six sites per tooth (mesio, mid, and distobuccal, and mesio, mid, and distopalatal) using a Williams periodontal probe (Nordent Manufacturing Inc., Elk Grove Village, IL, USA) calibrated in millimeters.

The patients were instructed to record the postoperative degrees of pain, redness, swelling, and functional complications, including chewing and speech, on a 10 cm horizontal visual analog scale (VAS), by placing a vertical mark between the two endpoints, from the first through seventh days. The scale was graded from left to right with values ranging from "0" (no pain, functional complications, discomfort, swelling, or redness) to "10" (worst pain, extreme functional complications, extreme discomfort, extreme swelling, and extreme redness). The keratinized gingiva width (KGW), attached gingiva width (AGW), and attached gingiva thickness (AGT) were also recorded before the surgery. Postoperative analyses were performed at four separate times: immediately, at the first week, and at the first and third months after surgery. The patients in each group were also asked if they required anesthesia during the operation and analgesics after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Those subjects with maxillary anterior frenula extending to the interdental papilla of the central incisors, those undergoing frenectomies for orthodontic, prosthodontic, or periodontal treatment and those with no surgical contraindications were included in this study.

Exclusion Criteria:

* The patients were excluded if they exhibited poor oral hygiene, received periodontal therapy, were being treated with antibiotics, anti-inflammatories, or analgesics during the previous three months, or if they had any systemic conditions that could affect oral surgery.

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
postoperative degrees of pain | Change from postoperative first week at postoperative third month
  visual analog scale (0 to 10 cm)

SECONDARY OUTCOMES:
plague index | preoperative
  between 0 to 4 scale
functional complications | Change from postoperative first week at postoperative third month
  visual analog scale (0 to 10 cm)

CONTACTS AND LOCATIONS:
Overall Officials: Ahu Uraz, PhD Dr, Study Director — Gazi University Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No
The patients will be instructed to record the postoperative degrees of pain, redness, swelling, and functional complications, including chewing and speech, on a 10 cm horizontal visual analog scale (VAS), by placing a vertical mark between the two endpoints, from the first through seventh days.

REFERENCES:
- [Background] Vescovi P, Corcione L, Meleti M, Merigo E, Fornaini C, Manfredi M, Bonanini M, Govoni P, Rocca JP, Nammour S. Nd:YAG laser versus traditional scalpel. A preliminary histological analysis of specimens from the human oral mucosa. Lasers Med Sci. 2010 Sep;25(5):685-91. doi: 10.1007/s10103-010-0770-4. PMID 20393771
- [Background] Fornaini C, Rocca JP, Bertrand MF, Merigo E, Nammour S, Vescovi P. Nd:YAG and diode laser in the surgical management of soft tissues related to orthodontic treatment. Photomed Laser Surg. 2007 Oct;25(5):381-92. doi: 10.1089/pho.2006.2068. PMID 17975951
- [Background] Romanos G, Nentwig GH. Diode laser (980 nm) in oral and maxillofacial surgical procedures: clinical observations based on clinical applications. J Clin Laser Med Surg. 1999 Oct;17(5):193-7. doi: 10.1089/clm.1999.17.193. PMID 11199822